CLINICAL TRIAL: NCT06030219
Title: Microbiome Effect of Omadacycline on Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Principal Investigator, Kevin W. Garey, Professor and Chair, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: G0505124
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: omadacycline; microbiome; healthy volunteer
MeSH Terms: interventions — omadacycline; Vancomycin; Moxifloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Omadacycline (Experimental): Subjects will receive 3 tablets on day 1 and day 2 (450 mg) followed by 2 tablets (300 mg) for days 3 through 10.
  Interventions: Drug: Omadacycline
- Vancomycin (oral) (Active Comparator): Vancomycin 125 mg capsules will be taken four times daily for a total of 10 days.
  Interventions: Drug: Vancomycin Pill
- Moxifloxacin (Active Comparator): Moxifloxacin 400 mg tablets will be taken once per day for a total of 10 days.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Omadacycline — 10-day course
  Arms: Omadacycline
Drug: Vancomycin Pill — 10-day course
  Arms: Vancomycin (oral)
Drug: Moxifloxacin — 10-day course
  Arms: Moxifloxacin

SUMMARY:
The goal of this study is to assess microbiome changes associated with omadacycline vs. comparators (moxifloxacin or oral vancomycin). Using a phase I study design, healthy volunteers aged 18-40 years will be given a 10-day course of either omadacycline 450 mg days 1 and 2 followed by 300 mg PO once daily, moxifloxacin 400 mg once daily, or oral vancomycin 125 mg given four times daily. Stool will be collected at baseline, daily during therapy, and at two follow-up time periods (days 13-14 and days 30-32). DNA will be extracted from stool and used for qPCR biomass and microbial metagenomic experiments. Results from the study will provide definitive data on the microbiome effects of omadacycline versus comparator antibiotics.

ELIGIBILITY:
Inclusion. All volunteers will be considered healthy based on medical history

Exclusion. Patients will be excluded if they report any of the following:

* Cardiovascular disease
* Gastrointestinal disease
* Hepatic or renal disease
* Receipt of an antibiotic for at least three months prior to enrollment.
* Receipt of a probiotic for at least a month prior to enrollment and during the entire study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Microbiome changes | During dosing and 30 day follow up period
  Metagenomic changes (16S rRNA) and qPCR for individual bacterial species

CONTACTS AND LOCATIONS:
Overall Officials: Kevin W Garey, Principal Investigator — Professor and Chair
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Metagenomic and metadata will be shared by posting to relevant biorepositories or upon reasonable requests from external investigators.

REFERENCES:
- [Derived] Ayele H, Jo J, Begum K, Hu C, Le TM, Alam MJ, Eubank TA, Haidacher SJ, Horvath TD, Hanson BM, Garey KW. A Randomized Phase 1 Study Investigating Gut Microbiome Changes With Moxifloxacin vs Oral Vancomycin: Implications for Clostridioides difficile Risk. J Infect Dis. 2025 Dec 20;232(6):1446-1456. doi: 10.1093/infdis/jiaf512. PMID 41081530
- [Derived] Jo J, Hu C, Horvath TD, Haidacher SJ, Begum K, Alam MJ, Garey KW. Phase I trial comparing bile acid and short-chain fatty acid alterations in stool collected from human subjects treated with omadacycline or vancomycin. Antimicrob Agents Chemother. 2025 Feb 13;69(2):e0125124. doi: 10.1128/aac.01251-24. Epub 2025 Jan 17. PMID 39819014
- [Derived] Jo J, Hu C, Begum K, Wang W, Le TM, Agyapong S, Hanson BM, Ayele H, Lancaster C, Jahangir Alam M, Gonzales-Luna AJ, Garey KW. Fecal Pharmacokinetics and Gut Microbiome Effects of Oral Omadacycline Versus Vancomycin in Healthy Volunteers. J Infect Dis. 2024 Jan 12;229(1):273-281. doi: 10.1093/infdis/jiad537. PMID 38051631

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT06030219/Prot_SAP_000.pdf